CLINICAL TRIAL: NCT02383420
Title: Clinical Evaluation of the Carestream PRO 3543 and PRO 3543C Digital Detectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 6M2375
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Predicate & Invest-GOS (Experimental): Radiation - Each subject will receive one x-ray using the predicate detector and one x-ray using the GOS investigational detector.
  Interventions: Radiation: Radiation
- Predicate & Invest-CsI (Experimental): Radiation - Each subject will receive one x-ray using the predicate detector and one x-ray using the CsI investigational detector.
  Interventions: Radiation: Radiation
- Predicate & Invest.-Cadavers GOS & CsI (Experimental): Radiation - Multiple exams (head, chest, legs, etc) were made on the cadavers. Each exam area received one x-ray using the predicate detector and two x-rays using both the GoS and the CsI investigational detector.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Live subjects will receive two x-rays, one with predicate detector and one using the GOS or CsI investigational detector. Multiple exams (head, chest, legs, etc) were made on the cadavers. Each exam area received one x-ray using the predicate detector and two x-rays using both the GoS and the CsI investigational detector.

SUMMARY:
The purpose of this clinical study is to evaluate the imaging performance of the Carestream PRO 3543 Detector and Carestream PRO 3543C Detector (referred to as the "investigational devices") as compared to the currently marketed Carestream DRX-1 Detector (referred to as the "predicate device"). Both detectors are flat panel digital imaging devices. The results of this study will be included in a Traditional 510(k) FDA Submission to obtain clearance to market the new detectors in the US. The study was designed in accordance with the FDA Guidance titled "Guidance for the Submission of 510(k)'s for Solid State X-ray Imaging Devices", issued on August 6, 1999.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the imaging performance of the investigational devices as compared to the currently marketed predicate device. The evaluation will consist primarily of comparing the diagnostic image quality of pediatric and adult cadaver studies and adult live human subject studies acquired under the same exposure technique.

Under the same position and radiological technique, pediatric and adult cadaver studies, and adult live human subject studies, using double-exposed images will be acquired to evaluate the diagnostic image quality of the investigational device versus the predicate device. Target images will be assembled and reviewed in a side-by-side Comparative Evaluation to statistically confirm the findings of this evaluation.

The live human subject portion of this study will be performed on healthy volunteers. Each volunteer will sign an Informed Consent after which they will have two (2) x-rays taken.The first x-ray will follow standard technique using the cleared predicate detector currently in use at the site. Following the first x-ray, we will take one additional x-ray of the same part of the body with one (1) of the investigational detectors. The x-ray from the investigational detector will not be used to diagnose.

If the x-ray obtained by the standard DR x-ray detector shows any unforeseen, unusual or abnormal findings, these findings will be communicated to the subject and their doctor by USPS mail.

Reason for Observational Study Type: There are three (3) physical detectors being used in this study. Each detector is 35 centimeters by 43 centimeters. None of the subjects will given a detector. All subjects are healthy volunteers recruited by flyer. All subjects will be imaged with the same predicate detector and one (1) of the investigational detectors.

ELIGIBILITY:
Inclusion Criteria:

* X-ray images of nearly identical positioning and exposure
* No visible image artifacts
* Subject 21 years or older
* Subject has provided informed consent
* Subject is in good general health (is able to be still to reduce the potential of motion in the images)
* Subject is able to stand for two (2) x-rays

Exclusion Criteria:

* Images that are not clinically acceptable for clinical radiographic reading as determined by the Principal Investigator.
* Subject is pregnant or suspicious of being pregnant
* Subject not able or willing to provide Informed Consent, or consent is withdrawn
* Not able to collect all required case information
* Subject has a history of high radiation exposure:
* Subject has undergone radiation therapy
* Subject has had two (2) or more CT scans within the past year

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hobbs, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Predicate & Invest.-GOS: Each subject will receive one x-ray using the predicate detector and one x-ray using the GOS investigational detector.
- Predicate & Invest.-CsI: Each subject will receive one x-ray using the predicate detector and one x-ray using the CsI investigational detector.
- Predicate & Investigational-Cadavers: Radiation - Multiple exams (head, chest, legs, etc) were made on the cadavers. Each exam area received one x-ray using the predicate detector and two x-rays using both the GoS and the CsI investigational detector.
Period: Overall Study
Arm/Group | Predicate & Invest.-GOS | Predicate & Invest.-CsI | Predicate & Investigational-Cadavers
Started | 10 | 10 | 3
Completed | 8 | 10 | 3
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Predicate & Invest.-CsI: Radiation - Each subject will receive one x-ray using the predicate detector and one x-ray using the CsI investigational detector.
- Total: Total of all reporting groups
Arm/Group | Predicate & Invest.-GOS | Predicate & Invest.-CsI | Predicate & Invest.-Cadavers GOS & CsI | Total
Number analyzed (Participants) | 8 | 10 | 3 | 21
Age, Customized [Number; unit: participants]
  21 years and older | 8 | 10 | 3 | 21
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 8 | 10 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Radlex Scale for Diagnostic Capability Ratings
Description: 1-Non-diagnostic Unacceptable for diagnostic purposes. Little or no clinically usable diagnostic information (e.g., gross underexposure, system failure or extensive motion artifact). Almost all such imaging should be repeated. 2-Limited Acceptable, with some technical defect (motion artifact, body habitus/poor x-ray penetration, or patient positioning may limit visualization of some body-regions but still adequate for diagnostic purposes). Not as much diagnostic information as is typical for an examination of this type, but likely sufficient. 3-Diagnostic Image quality that would be expected routinely when imaging cooperative patients. 4-Exemplary Good, most adequate for diagnostic purposes. Image quality that can serve as an example that should be emulated.
Time Frame: 9 weeks after last x-ray capture
Population: A total of 177 image pairs were included for the reader study. Of the 177 pairs, 160 were cadaver image pairs. A total of seventeen (17) adult live human subject pairs were included in the reader study.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Groups:
- Predicate: DRX-1 Detector, Live Subjects and Cadavers
- Investigational: DRX PRO 3543/C (GOS & CsI) Detectors, Live Subjects & Cadavers
Arm/Group | Predicate | Investigational
Number analyzed (Participants) | 20 | 20
Number analyzed (images) | 177 | 177
units on a scale | 3.0610 (0.0140) | 3.0633 (0.0141)
Statistical Analysis 1: Comparison: Predicate vs Investigational; Test type: Superiority or Other; p = 0.415, t-test, 2 sided — Level of significance (alpha) = 0.05

2. Secondary Outcome: Pair Preference Rating Scale
Description: During the Reader Study the radiologists completed a paired preference rating using the following scale: -3, Image displayed on left is strongly preferred; -2, Image displayed on left is moderately preferred; -1, Image displayed on left is slightly preferred; 0, No preference between the images; 1, Image displayed on right is slightly preferred; 2, Image displayed on right is moderately preferred; 3, Image displayed on right is strongly preferred. Both the predicate and investigational images were randomly assigned to appear on the right or left monitors. A spreadsheet was used for managing the data. Prior to analysis, raw ratings were converted so that those in favor of the investigational device were made positive, and ratings in favor of the predicate device were made negative.
Time Frame: 9 weeks after last x-ray capture
Population: cadavers and live human subjects
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: units
Groups:
- Image Pair Preference: Preference for predicate detector DRX-1 image versus preference for investigational DRX-PRO 3543/C (GOS & CsI) and vice versa.
Arm/Group | Image Pair Preference
Number analyzed (Participants) | 20
Number analyzed (units) | 177
units on a scale | 0.1333 (0.0209)
Statistical Analysis 1: Comparison: Image Pair Preference; Test type: Superiority or Other; p = 0.0000, t-test, 1 sided — Level of significance (alpha) = 0.05

ADVERSE EVENTS:
Time Frame: AE's were monitored for one month, March 2015.
Groups:
- Predicate & Invest.-Cadavers GOS & CsI: Multiple exams (head, chest, legs, etc) were made on the cadavers. Each exam area received one x-ray using the predicate detector and two x-rays using both the GoS and the CsI investigational detectors.
Arm/Group | Predicate & Invest.-GOS | Predicate & Invest.-CsI | Predicate & Invest.-Cadavers GOS & CsI
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No